CLINICAL TRIAL: NCT01804725
Title: Phase 1: To Compare Perineal Artery Occlusion in Road and Stationary Models. Phase 2: To Test Different Seats for Perineal Arterial Occlusion.
Brief Title: Study of Bicycle Seat Effects on Male Perineal Blood Flow
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Dr. Craig Niederberger, Clarence C. Saelhof Professor and Head, University of Illinois at Chicago
Other Study IDs: 2007-0284
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Effect of Bike Seats on Male Perineal Blood Flow
Keywords: bike seats; Erectile dysfunction; Perineum; Impotence
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective is to study the effects of bicycle riding and bicycle seats on blood flow to a man's reproductive organs. It has been shown that bicycle riding can affect a man's ability to have an erection. Each year, newer and better bicycle seats come out but these seats have not been adequately studied for their effects on blood flow in the genital region.

DETAILED DESCRIPTION:
Introduction:

An independent market research company released a report in 1997, estimating the bicycling industry to be worth an astounding 4.5 billion dollars.(1) The magnitude of this number gives us an idea of the popularity of this sport. An important component of a bicycle is its saddle, which can affect comfort, performance, and the rider's health. Several studies have reported sexual side effects in male bicyclists, more specifically temporary genital numbness and erectile dysfunction. Goldstein et. al claimed in their article that prolonged pressure on the perineal region causes arterial damage resulting in erectile dysfunction in men. These results have triggered bike manufacturers to come up with various saddle designs that claim to reduce risks for men. For this project investigators want to correlate bike riding and its effects on the male reproductive organs by measuring the pressures exerted on the perineum and blood flow while cycling. Previous studies on this matter have shown that a higher percentage of bicyclists are effected by Erectile Dysfunction(ED) compared to the general population. There are many published studies on the hemodynamics of the penis using Pulse Oximetry, Doppler Ultrasound and CAPSV measurements. Investigators goal is to be able to measure the pressures exerted on the arteries supplying the penis via the saddle over the perineum. A study, which attempted to carry out a measurement similar to this, used pressure transducers placed on the saddle of a stationary bike. There are flaws in this study, which investigators want to improve upon in designing this research experiment. For example, placing the sensors on the saddle enables measurements of force on the saddle and does not directly relate to the pressures exerted on the perineum. In other words by placing the sensors on the saddle researchers will not be able to distinguish between the pressures exerted on the perineum and other body parts in contact with the sensors on the seat, such as the sit bones. Also, while using a stationary bike the physics of the body and forces on the perineum are very different compared to road bikes on the road and mountain bikes on rough terrain. Investigators study corrects these flaws.

Purpose of study:

Can investigators measure the blood flow to the perineum via the perineal arteries and see the effect of bicycle riding on the blood flow through these arteries?

Design:

This is a pilot study which involved 2 steps to determine perineal blood flow and how bicycle seats affect this flow. The first step will be to use doppler ultrasound to measure the perineal blood flow in the Ultrasound suite of the University Illinois Chicago Medical Center. At this visit, patients will be asked to lie down in a frog-leg/lithotomy position on an exam table to allow access to the perineum. The linear ultrasound probe (L12-55) will be used to measure the flow through the perineal/cavernosal arteries. By applying sequentially increasing pressure, the critical pressure for occlusion will be measured along with flow rates at various applied perineal pressures. The second step will involve a bicycle ride where perineal pressures will be measured. Investigators use disposable sensors and tegaderm to stick the sensors on the perineum. No shaving of the perineum will be required so long as the sensor is able to be secured. The recording device is credit card size and will attach to the bicycle. The subjects ride using six different bike seats in a standard road course and also on a stationary trainer. This will conclude the requirement of the patient. The pressures obtained on the bicycle ride will be compared to the critical occlusion pressures and flow-pressure relationships measured in the ultrasound suite.

Recruitment:

Patients will be recruited for the project via various bicycle meetings. Cyclist will be approached via oral presentation and they will be men between ages 18-64, avid cyclists and will not be at risk of undue influence (i.e. UIC students). Please see attached recruitment script.

Risks Involved:

The study involves minimal risk to the subject as the subject will already be a cyclist and will be used to the mild exercise involved of cycling. Sensors will not use any electric input and the patient is at no harm from them. All data will be acquired using noninvasive radiology, ultrasound with doppler.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 18-64 male

Exclusion Criteria:

* none

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers will be recruited from the general population. Recruitment will be done using oral presentation, meetings, advertisement flyers.Participants will be avid cyclists and will not be at risk of undue influence( i.e UIC students).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-08; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Arteries occluding time for each seat | two years
  This measure indicates the time period the subjects are occluding their blood vessels in the perineal region. Different seats can occlude the arteries for different duration. So this measure tells us exactly what is the impact of each tested seat on male perineal blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Craig S Niederberger, M.D, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States